CLINICAL TRIAL: NCT01537874
Title: MassCONECT 4 Kids: Promoting Smoke-free Homes MassCONECT (Massachusetts Community Networks to Eliminate Cancer Disparities Through Education)
Brief Title: MassCONECT (Massachusetts Community Networks to Eliminate Cancer Disparities Through Education) 4 Kids: Promoting Smoke-free Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Vaughan Rees, Lecturer, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R24MD002772 (NIH); R24MD002772 (NIH)
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Tobacco Smoking Behavior
Keywords: Secondhand smoke; Pediatric disease
MeSH Terms: conditions — Smoking | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interview Intervention (Experimental): Motivational interviewing session (1 hour in home) plus 2 follow-up phone calls
  Interventions: Behavioral: Motivational Interview
- Usual Best Practices (Other): Standard care delivered using informational materials
  Interventions: Behavioral: Usual best practices

INTERVENTIONS:
Behavioral: Motivational Interview — 30 - 45 minutes in-person session to deliver results of nicotine air monitor and discuss home smoking ban using motivational interview techniques
  Arms: Motivational Interview Intervention
Behavioral: Usual best practices — Standard care delivered using informational materials
  Arms: Usual Best Practices

SUMMARY:
This study evaluates the effectiveness of a motivational interviewing intervention with families with young children ages 0-5 where smoking is happening in the home to adopt a smoke-free home plan and reduce child's second-hand smoke exposure.

DETAILED DESCRIPTION:
Involuntary secondhand smoke (SHS) exposure in homes is an entirely preventable public health threat that disproportionately burdens young children in communities of low socioeconomic position. Breathe Free For Kids is a community-based participatory research (CBPR) initiative to evaluate the effectiveness of Ml compared with usual best practices (UBP) by having parents voluntarily adopt smoke-free home policies to protect children from SHS. The Motivational Interviewing intervention protocol was developed in conjunction with community partners, integrated into a health department-sponsored home visiting program for high-risk children and other community-based agencies serving children, and delivered by trained community health workers.

ELIGIBILITY:
Inclusion Criteria:

* Tobacco smoking occurs regularly (smoke a minimum of one cigarette/cigar per day or five cigarettes/cigars per week) inside the home or in an attached patio/porch, hallway or stairwell
* Primary caregiver of child aged birth to 5 years old (inclusive) enrolled in Massachusetts Early Intervention program, Healthy Families program or the general population in Boston, Lawrence and Worcester areas.
* Ability of a custodial parent aged 17 or older/legally authorized representative or primary caregiver of child enrolled in participating programs to give permission for the index child to provide saliva sample.
* Participant has access to a telephone to schedule study contacts and participate in follow-up calls

Exclusion Criteria:

* Not able to understand English or Spanish at a 8th grade level or above
* In poor physical or psychological health (self-reported and observed by Community Health Worker), for whom participating in this intervention study might compromise the child's or participant's welfare, or be impracticable
* Index child is a ward of the state

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2010-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Voluntary adoption of a home smoking ban | 6 Months

SECONDARY OUTCOMES:
Self-reported smoking in the home | 6 Months
Household nicotine concentrations | 6 Months
Child salivary cotinine | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Vaughan Rees, PhD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (3):
- United States (3):
  - Boston Alliance for Community Health, Boston, Massachusetts
  - City of Lawrence Mayor's Health Task Force, Lawrence, Massachusetts
  - Common Pathways, Worcester, Massachusetts

REFERENCES:
- [Background] Keske RR, Rees VW, Behm I, Wadler BM, Geller AC. Second-hand smoke exposure and mitigation strategies among home visitation workers. Tob Control. 2013 Jul;22(4):250-4. doi: 10.1136/tobaccocontrol-2011-050133. Epub 2011 Dec 18. PMID 22184207